CLINICAL TRIAL: NCT06807268
Title: A 16-WEEK, MULTICENTER, INTERVENTIONAL, PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO INVESTIGATE EFFICACY AND SAFETY OF ABROCITINIB IN CHILDREN 6 TO LESS THAN 12 YEARS OF AGE WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS
Brief Title: A Study of the Medicine Called Abrocitinib in Children 6 to Less Than 12 Years of Age With Moderate-to-Severe Eczema
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7451023; 2023-509121-51-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Eczema
Keywords: Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Abrocitinib (Experimental): Abrocitinib administered as liquid oral suspension.
  Interventions: Drug: Abrocitinib
- Matching Placebo (Placebo Comparator): Placebo administered as liquid oral suspension.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Abrocitinib — Abrocitinib administered as liquid oral suspension.
  Other Names: PF-04965842
  Arms: Abrocitinib
Other: Placebo — Placebo administered as liquid oral suspension.
  Arms: Matching Placebo

SUMMARY:
This research study is being conducted to find out if the test medicine, abrocitinib, improves eczema and is safe for children 6 to <12 years of age who have moderate-to-severe eczema. Research study participants who meet the study criteria will be assigned by chance (like the flip of a coin) to receive either abrocitinib test medicine or placebo (pretend medicine that looks just like the test medicine) for 16 weeks. The study will last for about 24 weeks in total.

DETAILED DESCRIPTION:
Different questionnaires will be used to find out how the participant's eczema is doing during the research study. An electronic diary, which looks like a cellular phone, will be used to collect the questionnaire information and other research study-related information. It will also be used to remind participants to take the test medicine each day and to fill out the questionnaires. Participants will also be asked to wear something on their wrist that looks like a children's wristwatch so we can know when they are scratching their skin because of their atopic dermatitis. Laboratory tests, physical examinations and vital signs (height, weight, temperature, blood pressure and heart rate) will be conducted before and during the research study to monitor your child's health. Participants will need to come to the clinic for research study visits and at other times during the research study, the research study doctor or nurse will call the participants to find out the participant is doing.

ELIGIBILITY:
Inclusion Criteria Children aged 6 to <12 years at the time of informed consent/assent.

• No contraception methods are required for male participants. Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

Disease Characteristics:

Participants who meet all of the following AD criteria:

* A documented diagnosis of chronic AD for at least 1 year prior to screening and confirmed at screening and baseline visits according to the Hanifin and Rajka criteria[19]; and
* A diagnosis of moderate-to-severe AD at the baseline visit (must fulfill all of the following criteria: BSA ≥10%, vIGA ≥3, EASI ≥16, and WI-NRS ≥4); and
* Documented history (within 6 months of the screening visit) of inadequate response to treatment with topical medical therapy for AD (eg, TCS and TCI), for at least 4 weeks and are candidates for systemic therapy

Other Inclusion Criteria:

Body weight ≥15 kg

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

If the participant has SDQ total score ≥17, the investigator should exclude them or refer the child to a pediatric MHP to determine if it is safe to participate in the study. A copy or summary of the evaluation should be placed in the site source documents.

Have any of the following medical conditions:

* Infections:

  * Skin infections that require treatment with systemic antimicrobials within 2 weeks prior to Day 1 (Baseline) or have superficial skin infections within 1 week of Day 1.
  * History of systemic infection requiring hospitalization or parenteral antimicrobial therapy or as otherwise judged clinically significant by the investigator within 1 month prior to Day 1.
  * Have a history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent localized, dermatomal herpes zoster.
  * Infection with HIV, hepatitis B, and/or hepatitis C
  * Evidence of active TB or inadequately treated latent TB.
* Skin Conditions:

  - Including but not limited to psoriasis, seborrheic dermatitis or lupus on Day 1 that would interfere with evaluation of AD or response to treatment.
* Other Conditions:

  * Documented history of skeletal dysplasia.
  * Documented history of retinal detachment.
  * History of or conditions associated with thrombocytopenia, coagulopathy or platelet dysfunction.
  * Prior history of leukemia, lymphoma, sarcoma or any other malignancy.
  * Immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.
  * Any other medical conditions that in the investigator's judgment make the participant inappropriate for the study.

Prior/Concomitant Therapy:

Prior treatment with a systemic JAK inhibitor for AD. Live attenuated vaccination within 6 weeks prior to Day 1 or require vaccination with live attenuated vaccines during treatment or within 6 weeks after the last dose of study intervention.

Concomitant use of strong inhibitors and inducers of CYP2C19 enzymes, strong inducers of CYP2C9 enzymes, P-gp substrates with narrow therapeutic index and sensitive CYP2C19 substrates is not allowed in the study.

Prior/Concurrent Clinical Study Experience:

Previous administration of an investigational drug within 30 days or 5 half lives, whichever is longer, of Day 1.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Response based on achieving Validated Investigator's Global Assessment (vIGA) score of clear (0) or almost clear (1) (on a 5-point scale) and a reduction from baseline of ≥2 points at Week 12 | At week 12
  The difference in proportion of responders based on vIGA at Week 12 in patients with moderate-to-severe AD treated with abrocitinib versus placebo
Response based on achieving ≥75% improvement from baseline in the Eczema Area and Severity Index (EASI)-75 at Week 12 | At week 12
  The difference in proportion of responders based on EASI-75 at Week 12 in patients with moderate-to-severe AD treated with abrocitinib versus placebo

SECONDARY OUTCOMES:
Change from Baseline (CFB) in the Worst Itch Numerical Rating Scale (WI-NRS) at Week 2 | At week 2
  The difference in mean CFB in WI-NRS total score at Week 2 in patients with moderate-to-severe AD treated with abrocitinib versus placebo
Response based on achieving at least a 4-point improvement from baseline in the WI-NRS at Week 12 | At week 12
  The difference in proportion of responders based on achieving at least a 4-point improvement from baseline in the WI-NRS at Week 12 in patients with moderate-to-severe AD treated with abrocitinib versus placebo
Response based on achieving WI-NRS <2 at Week 12 | At week 12
  The difference in proportion of responders based on achieving WI-NRS <2 at Week 12 in patients with moderate-to-severe AD treated with abrocitinib versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (6):
  - Cahaba Dermatology & Skin Health Center, LLC, Birmingham, Alabama
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Tribe Clinical Research, LLC, Greenville, South Carolina
- China (5):
  - Beijing Children's hospital, Capital Medical University, Beijing, Beijing Municipality
  - Hunan Children's Hospital, Changsha, Hunan
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Xinhua Hospital Affiliated to Shanghai JiaoTong University School of Medicine, Shanghai
- Germany (2):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
- Hungary (2):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Clinexpert Kft., Budapest, Pest County
- Japan (5):
  - Queen's square Medical Facilities Queen's square Dermatology and Allergology, Yokohama, Kanagawa
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Sasamoto Children's Clinic, Setagaya-ku, Tokyo
  - Fukuoka National Hospital, Fukuoka
- Mexico (2):
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - Servicios Hospitalarios de Mexico S.A. DE C.V., Chihuahua City
- Poland (6):
  - LUXDERM Specjalistyczny Gabinet Dermatologiczny prof. dr hab. n. med. Dorota Krasowska, Lublin, Lublin Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - DERMAPOLIS Medical Dermatology Center dr n. med. Edyta Gebska, Chorzów, Silesian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Dermoklinika - Centrum Medyczne spółka cywilna M. Kierstan, J. Narbutt, A. Lesiak, Lodz, Łódź Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Spain (3):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital General de Granollers, Granollers, Barcelona [barcelona]
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451023